CLINICAL TRIAL: NCT07154407
Title: The Effectiveness of AI-assisted Masticatory Muscle Training on Oral Hygiene, Masticating, and Swallowing in Patients With Schizophrenia
Brief Title: AI-assisted Masticatory Muscle Training in Patients With Schizophrenia
Acronym: AI-assisted
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(I)-20240124
Record Dates: First submitted 2025-08-11; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia Disorder
Keywords: Masticatory Muscle Training; AI-assisted; Oral Hygiene; Masticate; Swallow
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervented group (Experimental): The group member (n=50) will receive 'AI-assisted Masticatory Muscle Training' sessions, each lasting 20 minutes, before each of their three daily meals. The plaque index, Winkle tongue-coating index, dry mouth, repetitive saliva swallowing, saliva flow rate, biting force, tongue pressure, oral frailty, RSST, DDK, and oral care behaviors were assessed at baseline, as well as during the 3-month and 6-month follow-ups.
  Interventions: Other: AI-assisted Mastisting Training App
- Controlled group (No Intervention): The control group (n=50) will be maintained their scheduled activities in daycare as usual. The plaque index, Winkle tongue-coating index, dry mouth, repetitive saliva swallowing, saliva flow rate, biting force, tongue pressure, oral frailty, RSST, DDK, and oral care behaviors were assessed at baseline, as well as during the 3-month and 6-month follow-ups.

INTERVENTIONS:
Other: AI-assisted Mastisting Training App — An artificial intelligence (AI) recognition system for the 'AI-assisted Masticatory Muscle Training,' tailored to train masticatory muscles in patients with schizophrenia. By finishing certain exercise per day, expecting the experimental oral hygience, masticating and swallowing fuction could be advanced,
  Arms: Intervented group

SUMMARY:
Dysphagia seems to be quite common and potentially severe in schizophrenia, which may lead to acute asphyxia or pneumonia. Dysphagia in schizophrenia could be associated with drug-induced Parkinsonism, dystonia, tardive dyskinesia, dry mouth, excessive saliva, and other complications. Inadequate oral hygiene may lead to the accumulation of plaque, which can cause oral diseases and consequently result in tooth loss. This could be one of the significant factors affecting impaired masticating and swallowing abilities.

An experimental study with random assignment will be adopted. The participants from 2 hospitals will be assigned to two groups: experimental group (n=50), and control group (n=50). The experimental group will receive 'AI-assisted Masticatory Muscle Training' sessions, each lasting 20 minutes, before each of their three daily meals. The plaque index, Winkle tongue-coating index, dry mouth, repetitive saliva swallowing, saliva flow rate, biting force, tongue pressure, oral frailty, RSST, DDK, and oral care behaviors were assessed at baseline, as well as during the 3-month follow-ups.

DETAILED DESCRIPTION:
Dysphagia seems to be quite common and potentially severe in schizophrenia, which may lead to acute asphyxia or pneumonia. Dysphagia in schizophrenia could be associated with drug-induced Parkinsonism, dystonia, tardive dyskinesia, dry mouth, excessive saliva, and other complications. Inadequate oral hygiene may lead to the accumulation of plaque, which can cause oral diseases and consequently result in tooth loss. This could be one of the significant factors affecting impaired masticating and swallowing abilities.

An experimental study with random assignment will be adopted. The participants from 2 hospitals will be assigned to two groups: experimental group (n=50), and control group (n=50). The experimental group will receive 'AI-assisted Masticatory Muscle Training' sessions, each lasting 20 minutes, before each of their three daily meals. The control group will be maintained their scheduled activities in daycare as usual. The plaque index, Winkle tongue-coating index, dry mouth, repetitive saliva swallowing, saliva flow rate, biting force, tongue pressure, oral frailty, RSST, DDK, and oral care behaviors were assessed at baseline, as well as during the 3-month follow-ups. Generalized Estimating Equations (GEE) were used to analyses the indicated effects.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric Outpatient Ward Schizophrenia Diagnosed patient with 20 years or above
* Without Violence or suicidal tendencies
* With a self-owned smartphone
* Able to stabilise the IOPI machine while testing
* Able to communicate

Exclusion Criteria:

* Severe psychiatric symptoms
* With medical history which affects oral hygiene and masticating function severely (such as stroke, oral cavity-related cancer, periodontitis)
* Severe cognitive function with a score of less than 16 marks in the MoCA Test
* Indicated with Motor Neuron Disease
* Joining multiple Intervention Experiments simultaneously

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-11 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anterior tongue strength | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using the IPOI machine to test participants' tongue strength once a month for a total of 3 months, and a follow-up review 3 months after the end of treatment
Posterior tongue strength | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using the IPOI machine to test participants' tongue strength once a month for a total of 3 months, and a follow-up review 3 months after the end of treatment
Masticatory Performace | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using colour-changing chewing gum to assess the ability, the colour would be changed according to the frequency of chewing
Oral Hygiene | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using the Plaque index, Winkle tongue-coating index to assess participants' oral hygiene
Swallowing Performance | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using the Repetitive Saliva Swallowing Test to assess the ability to swallow. The times of participants swallowed within 30 seconds would be recorded
Oral Care Behaviours | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using a survey to collect participants' behaviours
Cognitive Function | From day 1 of enrollment to the end of the treatment period (up to 3 months)
  Using MoCA to assess cognitive ability once at the beginning of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh Hsiu Fen, PhD, Principal Investigator — Kaohsiung medical university nursing faculty

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT07154407/Prot_SAP_000.pdf